CLINICAL TRIAL: NCT02341417
Title: A Multicenter Single-arm Extension Study to Characterize the Long-term Safety of Cinacalcet Hydrochloride in the Treatment of Secondary Hyperparathyroidism in Pediatric Subjects With Chronic Kidney Disease on Dialysis
Brief Title: Extension Study of Cinacalcet for Treatment of Secondary Hyperparathyroidism (SHPT) in Pediatric Patients With Chronic Kidney Disease on Dialysis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20140159; 2014-003563-38 (EudraCT Number)
Record Dates: First submitted 2014-12-02; First posted 2015-01-19 (Estimated); Results first posted 2018-05-18 (Actual); Last update posted 2020-06-29 (Actual); Status verified 2020-06

CONDITIONS: Secondary Hyperparathyroidism, Chronic Kidney Disease
Keywords: Chronic Kidney Disease, Dialysis, Secondary Hyperparathyroidism, Pediatric
MeSH Terms: conditions — Hyperparathyroidism, Secondary; Renal Insufficiency, Chronic | interventions — Cinacalcet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cinacalcet (Experimental): Participants received cinacalcet daily for 24 weeks in this extension study. For participants who received standard of care (SOC) in parent study 20130356, the starting dose was 0.20 mg/kg/day. For participants who received SOC and cinacalcet in parent study 20130356 or 20110100 the starting dose was either the same as the last dose received in the parent study or 0.20 mg/kg/day if the last dose of cinacalcet in the parent study was received > 14 days before day 1 of this study.
  Dose adjustments and withholding were based on weekly assessments of ionized calcium as well as plasma intact parathyroid hormone (iPTH) and corrected serum calcium levels assessed monthly.
  Interventions: Drug: Cinacalcet

INTERVENTIONS:
Drug: Cinacalcet — Cinacalcet was provided as 5 mg capsules for sprinkling or as 30 mg film-coated tablets for swallowing. The protocol-specified doses were: 1, 2.5, 5, 7.5, 10, 15, 30, 60, 90, 120, and 180 mg.
  Other Names: Cinacalcet hydrochloride, Cinacalcet HCL, Sensipar®, Mimpara®

SUMMARY:
The primary objective of this study was to characterize the long-term safety and tolerability of cinacalcet in pediatric patients with chronic kidney disease (CKD) receiving dialysis.

DETAILED DESCRIPTION:
This extension study was designed to characterize the long-term safety and tolerability of cinacalcet in pediatric patients from Amgen Studies 20130356 (NCT02138838) and 20110100 (NCT01439867) who either had completed the parent study or were ongoing at the time an administrative decision was made to end the parent study. After enrolling into this study participants were administered cinacalcet for 28 weeks or until the time of renal transplant or parathyroidectomy, whichever occurred first. The treatment period was followed by a 4-week safety follow-up period.

ELIGIBILITY:
INCLUSION CRITERIA:

All subjects:

* Subject's legally acceptable representative has provided informed consent when the subject is legally too young to provide informed consent and the subject has provided written assent based on local regulations and/or guidelines prior to any Study 20140159 activities/procedures being initiated.
* Dialysate calcium concentration ≥ 2.5 mEq/L at day 1

All subjects with > 14 days between the last study visit in Study 20130356 or Study 20110100 and screening for Study 20140159:

* Subjects on anti-convulsant medication must be on a stable dose

All subjects from 20130356:

* Completed treatment through week 20 in the 20130356 study or on study at the time of Study 20130356 termination
* Dry weight ≥ 12.5 kg at day 1 of Study 20140159

Subjects Randomized to the 20130356 Standard of Care Arm Only:

* intact parathyroid hormone (iPTH) value ≥ 300 pg/mL (within 7 days of day 1 in Study 20140159)
* Corrected calcium value ≥ 8.8 mg/dL within 7 days of day 1 in Study 20140159

All Subjects from 20110100:

* Completed week 26 End of Study visit in the, 20110100 study or on study at the time of Study 20110100 termination
* Dry weight ≥ 7 kg at day 1 of Study 20140159

EXCLUSION CRITERIA:

General (studies 20130356 and 20110100):

* Currently receiving treatment in another investigational device or drug study, or less than 30 days since ending treatment on another investigational device or drug study(s), other than Amgen Studies 20130356 or 20110100.
* Other investigational procedures while participating in this study are excluded.
* Malignancy except non-melanoma skin cancers, cervical or breast ductal carcinoma in situ within the last 5 years.
* Subject has known sensitivity to any of the products to be administered during dosing.
* Subject likely to not be available to complete all protocol-required study visits or procedures, and/or to comply with all required study procedures (eg, electronic patient diary [ediary]) to the best of the subject and investigator's knowledge
* History or evidence of any other clinically significant disorder, condition or disease (with the exception of those outlined above) that, in the opinion of the investigator or Amgen physician, if consulted, would pose a risk to subject safety or interfere with the study evaluation, procedures, or completion.
* Subject previously has entered this study.
* If sexually active, subject is not willing to use acceptable contraception during treatment and for at least 9 days after the end of treatment.
* Subject is pregnant or breast feeding, or planning to become pregnant during the study or within 9 days after the end of treatment
* History of congenital long QT syndrome, second or third degree heart block, ventricular tachyarrythmias, or other conditions associated with prolonged QT interval
* A new onset of seizures or worsening of pre-existing seizure disorder

All Subjects with > 14 days between the last study visit in Study 20130356 or Study 20110100 and the screening visit in Study 20140159 will have the following exclusion criteria applied during screening and day 1:

* Unstable chronic heart failure defined as worsening pulmonary edema or other signs and symptoms as per investigator assessment during screening
* Received therapy with commercial cinacalcet after the last study visit in Study 20130356 or Study 20110100 before day 1 of Study 20140159
* Scheduled date for kidney transplantation from a known living donor that makes completion of the study unlikely
* Either new or recurrent cardiac ventricular arrhythmias requiring a change in treatment within 10 days prior to screening visit or day 1 of Study 20140159 screening
* Hepatic impairment indicated by elevated levels of hepatic transaminase or bilirubin (aspartate aminotransferase [AST] ≥ 1.5 × upper limit of normal [ULN] OR alanine aminotransferase [ALT] ≥ 1.5 × ULN OR total bilirubin ≥ 1 × ULN per institutional laboratory range) during screening

All Subjects - Day 1 Study Visit:

* Subject has an ongoing adverse event from Studies 20130356 or 20110100 that is considered related to investigational product and is ≥ Common Terminology Criteria for Adverse Events (CTCAE) (v 4.0) grade 3, and/or considered clinically significant in the opinion of the investigator
* Central laboratory values were not obtained/are not available at day 1 in Study 20140159
* Corrected QT Interval (QTc) > 500 ms, using Bazett's formula
* QTc ≥ 450 to ≤ 500 ms, using Bazett's formula, unless written permission to enroll is provided by the investigator after consultation with a pediatric cardiologist
* Use of grapefruit juice, herbal medications, CYP3A4 inhibitors (eg, erythromycin, clarithromycin, ketoconazole, itraconazole), or CYP2D6 substrates (eg, flecainide, propafenone, metoprolol, desipramine, nortriptyline, clomipramine)
* Use of concomitant medications that may prolong the QTc interval (eg, ondansetron, albuterol)

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 28 (Actual)
Dates: Start 2015-06-10 (Actual); Primary Completion 2017-03-15 (Actual); Study Completion 2017-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (33):
- United States (18):
  - Research Site, Los Angeles, California
  - Research Site, Tucker, Georgia
  - Research Site, Baltimore, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Minneapolis, Minnesota
  - Research Site, Jackson, Mississippi
  - Research Site, Kansas City, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, West Orange, New Jersey
  - Research Site, New York, New York
  - Research Site, Greenville, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Cleveland, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, Salt Lake City, Utah
- Research Site, Brussels, Belgium
- Research Site, Prague, Czechia
- Research Site, Paris, France
- Germany (3):
  - Research Site, Hanover
  - Research Site, Heidelberg
  - Research Site, Marburg
- Research Site, Athens, Greece
- Research Site, Szeged, Hungary
- Research Site, Genova, Italy
- Poland (2):
  - Research Site, Krakow
  - Research Site, Lodz
- Russia (3):
  - Research Site, Moscow
  - Research Site, Saint Petersburg
  - Research Site, Samara
- Research Site, Kyiv, Ukraine

REFERENCES:
- [Background] Warady BA, Ng E, Bloss L, Mo M, Schaefer F, Bacchetta J. Cinacalcet studies in pediatric subjects with secondary hyperparathyroidism receiving dialysis. Pediatr Nephrol. 2020 Sep;35(9):1679-1697. doi: 10.1007/s00467-020-04516-4. Epub 2020 May 4. PMID 32367309
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 16 centers in United States, Russian Federation, Ukraine, Belgium, Czech Republic, Greece, France, and Poland.
Pre-assignment Details: This extension study enrolled participants who completed one of the parent studies 20110100 (NCT01439867) or 20130356 (NCT02138838). Results are reported by treatment received in the parent study.
Groups:
- 20130356 SOC: Participants who received standard of care (SOC) in parent study 20130356 received cinacalcet daily for up to 28 weeks in this extension study. The starting dose was 0.20 mg/kg/day. Dose adjustments and withholding were based on weekly assessments of ionized calcium as well as plasma intact parathyroid hormone (iPTH) and corrected serum calcium levels assessed monthly.
- 20130356 SOC + Cinacalcet: Participants who received SOC and cinacalcet in parent study 20130356 received cinacalcet daily for up to 28 weeks in this extension study. The starting dose was either the same as the last dose received in the parent study or 0.20 mg/kg/day if the last dose of cinacalcet in the parent study was received > 14 days before day 1 of this study. Dose adjustments and withholding were based on weekly assessments of ionized calcium as well as plasma intact parathyroid hormone (iPTH) and corrected serum calcium levels assessed monthly.
- 20110100 SOC + Cinacalcet: Participants who received SOC and cinacalcet in parent study 2011100 received cinacalcet daily for up to 28 weeks in this extension study. The starting dose was either the same as the last dose received in the parent study or 0.20 mg/kg/day if the last dose of cinacalcet in the parent study was received > 14 days before day 1 of this study. Dose adjustments and withholding were based on weekly assessments of ionized calcium as well as plasma intact parathyroid hormone (iPTH) and corrected serum calcium levels assessed monthly.
Period: Overall Study
Arm/Group | 20130356 SOC | 20130356 SOC + Cinacalcet | 20110100 SOC + Cinacalcet
Started | 13 | 14 | 1
Completed | 11 | 12 | 0
Not Completed | 2 | 2 | 1
Not completed — Withdrawal by Subject | 0 | 2 | 0
Not completed — Decision by sponsor | 2 | 0 | 0
Not completed — Death | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 20130356 SOC | 20130356 SOC + Cinacalcet | 20110100 SOC + Cinacalcet | Total
Number analyzed (Participants) | 13 | 14 | 1 | 28
Age, Continuous [Median (Full Range); unit: years] | 14.0 [9 to 18] | 14.0 [7 to 17] | 2.0 [2 to 2] | 14.0 [2 to 18]
Age, Customized [Count of Participants; unit: Participants] — One participants in the 20130356 SOC group was 17 years old at the time of enrollment of parent study and had turned 18 at the time of enrollment of Study 20140159.
  Participants
    28 days to < 2 years | 0 | 0 | 0 | 0
    2 to < 6 years | 0 | 0 | 1 | 1
    6 to < 12 years | 4 | 6 | 0 | 10
    12 to ≤ 18 years | 9 | 8 | 0 | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 10 | 0 | 18
  Male | 5 | 4 | 1 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 12 | 14 | 1 | 27
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Black (or African American) | 1 | 4 | 0 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  White | 12 | 9 | 1 | 22
  Other | 0 | 1 | 0 | 1
Intact Parathyroid Hormone (iPTH) [Median (Inter-Quartile Range); unit: pg/mL] — Intact parathyroid hormone levels are reported for the extension study baseline and also for baseline relative to day 1 of cinacalcet treatment (equivalent to baseline of extension study for participants who received SOC alone in parent study 20130356; transferred from parent study for all other participants).
  pg/mL
    Extension study baseline | 1432.69 [800.19 to 1695.48] | 1001.35 [525.76 to 1292.08] | 907.74 [907.74 to 907.74] | 1047.41 [583.37 to 1530.03]
    Day 1 of cinacalcet treatment baseline | 1432.69 [800.19 to 1695.48] | 798.10 [622.36 to 1360.95] | 992.60 [992.60 to 992.60] | 980.56 [639.85 to 1530.03]
Corrected Total Serum Calcium [Median (Inter-Quartile Range); unit: mg/dL] — Total serum calcium was corrected using the following formula if the serum albumin was < 4 g/dL:
  Corrected total serum calcium (mg/dL) = measured total serum calcium (mg/dL) + 0.8 (4.0 - serum albumin (g/dL)) Corrected calcium levels are reported for the extension study baseline and also for baseline relative to day 1 of cinacalcet treatment (equivalent to baseline of extension study for participants who received SOC alone in parent study 20130356; transferred from parent study for all other participants).
  mg/dL
    Extension study baseline | 9.56 [9.40 to 10.00] | 9.93 [9.02 to 10.16] | 10.29 [10.29 to 10.29] | 9.80 [9.36 to 10.18]
    Day 1 of cinacalcet treatment baseline | 9.56 [9.40 to 10.00] | 9.86 [9.58 to 10.18] | 10.90 [10.90 to 10.90] | 9.80 [9.45 to 10.19]
Ionized Calcium [Median (Inter-Quartile Range); unit: mmol/L]
  Extension study baseline | 1.130 [1.110 to 1.230] | 1.145 [1.100 to 1.280] | 1.390 [1.390 to 1.390] | 1.140 [1.110 to 1.260]
  Day 1 of cinacalcet treatment baseline | 1.130 [1.110 to 1.230] | 1.225 [1.140 to 1.270] | 1.340 [1.340 to 1.340] | 1.215 [1.125 to 1.260]
Serum Phosphorus [Median (Inter-Quartile Range); unit: mg/dL] — Phosphorus levels are reported for the extension study baseline and also for baseline relative to day 1 of cinacalcet treatment (equivalent to baseline of extension study for participants who received SOC alone in parent study 20130356; transferred from parent study for all other participants).
  mg/dL
    Extension study baseline | 5.57 [4.86 to 6.19] | 6.05 [5.31 to 6.67] | 8.08 [8.08 to 8.08] | 5.85 [5.23 to 6.58]
    Day 1 of cinacalcet treatment baseline | 5.57 [4.86 to 6.19] | 5.75 [4.88 to 6.13] | 9.00 [9.00 to 9.00] | 5.74 [4.87 to 6.32]
Calcium Phosphorus Product (Ca x P) [Median (Inter-Quartile Range); unit: mg²/dL²]
  Extension study baseline | 54.42 [48.59 to 58.82] | 57.80 [50.94 to 65.65] | 82.28 [82.28 to 82.28] | 56.71 [50.11 to 65.06]
  Day 1 of cinacalcet treatment baseline | 54.42 [48.59 to 58.82] | 57.98 [47.47 to 62.25] | 98.90 [98.90 to 98.90] | 56.81 [48.03 to 62.24]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: Adverse events (AEs) were graded according to the Common Terminology Criteria for Adverse Events (CTCAE, v4.0). The investigator assessed whether the adverse event was possibly related to the study drug as indicated by a "yes" or "no" response to the question: Is there a reasonable possibility that the event may have been caused by the study drug?
Time Frame: From first dose of study drug in the extension study up to 4 weeks after the last dose; 32 weeks.
Population: All enrolled participants who received at least one dose of study drug in the extension study.
Measure: Count of Participants; unit: Participants
Arm/Group | 20130356 SOC | 20130356 SOC + Cinacalcet | 20110100 SOC + Cinacalcet
Number analyzed (Participants) | 13 | 14 | 1
Participants
  Any adverse event (AE) | 9 | 10 | 1
  AE Grade ≥ 2 | 2 | 7 | 1
  AE Grade ≥ 3 | 2 | 6 | 1
  AE Grade ≥ 4 | 0 | 0 | 1
  Serious adverse event (SAE) | 2 | 6 | 1
  AE leading to discontinuation of study drug | 0 | 0 | 0
  Fatal adverse events | 0 | 0 | 1
  Treatment-related adverse events (TRAE) | 5 | 4 | 0
  Treatment-related AE Grade ≥ 2 | 0 | 1 | 0
  Treatment-related AE Grade ≥ 3 | 0 | 0 | 0
  Treatment-related AE Grade ≥ 4 | 0 | 0 | 0
  Treatment-related serious adverse events | 0 | 0 | 0
  TRAE leading to discontinuation of study drug | 0 | 0 | 0
  Fatal treatment-related adverse events | 0 | 0 | 0

2. Secondary Outcome: Percentage of Participants Achieving ≥ 30% Reduction in iPTH From Baseline to Mean Value During Weeks 11 and 15
Description: This endpoint was analyzed in participants who received SOC only in parent study 20130356.
  Participants who had no iPTH values during weeks 11 or 15 were considered non-responders. Data collected more than 7 days after the last dose of study drug were excluded.
Time Frame: Baseline (defined as the mean values of samples collected during the screening period and day 1 pre-dose in the extension study) and weeks 11 and 15
Population: Enrolled participants from Study 20130356 who did not receive cinacalcet prior to day 1 of the extension study and had ≥ 1 assessment after day 1 of the extension study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 20130356 SOC
Number analyzed (Participants) | 13
percentage of participants | 30.8 [9.1 to 61.4]

3. Secondary Outcome: Percentage of Participants Achieving ≥ 30% Reduction in iPTH From Baseline to Mean Value During Weeks 23 and 28
Description: This endpoint was analyzed in participants who received SOC only in parent study 20130356.
  For participants who had no values during week 23 and 28, the mean of the last 2 available post-baseline values collected in the dose-titration phase was used. If only 1 post-baseline value was available, this single value was used. If no post-baseline value was available, the participant was considered a non-responder. Data collected more than 7 days after the last dose of study drug were excluded.
Time Frame: Extension study baseline and weeks 23 and 28
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 20130356 SOC
Number analyzed (Participants) | 13
percentage of participants | 23.1 [5.0 to 53.8]

4. Secondary Outcome: Percent Change From Baseline in iPTH to the Mean Value During Weeks 23 and 28
Description: This endpoint was analyzed in participants who received SOC only in parent study 20130356.
  For participants who had no values during week 23 and week 28, the mean of the last 2 available post-baseline values collected in the dose-titration phase was used. If only 1 post-baseline value was available, this single value was used. If no post-baseline value was available, the participant was excluded from the analysis. Data collected more than 7 days after the last dose of study drug were excluded.
Time Frame: Extension study baseline and weeks 23 and 28
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | 20130356 SOC
Number analyzed (Participants) | 13
percent change | 11.43 [-20.64 to 27.27]

5. Secondary Outcome: Percentage of Participants Who Achieved Mean iPTH ≤ 300 pg/mL During Weeks 23 and 28
Description: For participants who had no values during week 23 and 28, the mean of the last 2 available post-baseline values collected in the dose-titration phase was used. If only 1 post-baseline value was available, this single value was used. If no post-baseline value was available, the participant was considered a non-responder. Data collected more than 7 days after the last dose of study drug were excluded.
Time Frame: Weeks 23 and 28
Population: All enrolled participants in the extension study (Study 20140159) who received at least one dose of cinacalcet during the extension study and had at least one assessment after day 1 of the extension study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 20130356 SOC | 20130356 SOC + Cinacalcet | 20110100 SOC + Cinacalcet
Number analyzed (Participants) | 13 | 14 | 1
percentage of participants | 7.7 [0.2 to 36.0] | 21.4 [4.7 to 50.8] | 0.0 [0.0 to 97.5]

6. Secondary Outcome: Change From Baseline in Corrected Serum Calcium to the Mean Value During Weeks 23 to 28
Description: For participants who had no values during weeks 23 to 28, the mean of the last 2 available post-baseline values collected in the dose-titration phase was used. If only 1 post-baseline value was available, this single value was used. If no post-baseline value was available, the participant was excluded from the analysis. Data collected more than 7 days after the last dose of study drug were excluded.
Time Frame: Extension study baseline and weeks 23 and 28
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | 20130356 SOC | 20130356 SOC + Cinacalcet | 20110100 SOC + Cinacalcet
Number analyzed (Participants) | 13 | 14 | 1
mg/dL | -0.24 [-0.46 to -0.06] | -0.24 [-0.81 to 0.58] | -0.74 [-0.74 to -0.74]

7. Secondary Outcome: Change From Baseline in Serum Phosphorus to the Mean Value During Weeks 23 to 28
Description: as for outcome 6
Time Frame: Extension study baseline and weeks 23 and 28
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | 20130356 SOC | 20130356 SOC + Cinacalcet | 20110100 SOC + Cinacalcet
Number analyzed (Participants) | 13 | 14 | 1
mg/dL | 0.19 [-0.52 to 0.56] | -0.08 [-1.41 to 0.17] | 0.82 [0.82 to 0.82]

8. Secondary Outcome: Serum Corrected Calcium at Baseline, Week 11, and Week 28
Description: Data collected more than 7 days after the last dose of study drug were excluded.
Time Frame: Extension study baseline, week 11 and week 28
Population: All enrolled participants in the extension study (Study 20140159) who received at least one dose of cinacalcet during the extension study and had at least one assessment after day 1 of the extension study, with available data at each time point.
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | 20130356 SOC | 20130356 SOC + Cinacalcet | 20110100 SOC + Cinacalcet
Number analyzed (Participants) | 13 | 14 | 1
mg/dL
  Extension study baseline | 9.56 [9.40 to 10.00] | 9.93 [9.02 to 10.16] | 10.29 [10.29 to 10.29]
  Week 11: number analyzed (Participants) | 12 | 12 | 0
  Week 11 | 9.35 [9.20 to 9.60] | 9.85 [9.30 to 10.65] |
  Week 28: number analyzed (Participants) | 9 | 12 | 0
  Week 28 | 9.50 [9.30 to 10.00] | 9.90 [9.10 to 10.25] |

9. Secondary Outcome: Serum Phosphorus at Baseline, Week 11, and Week 28
Description: Data collected more than 7 days after the last dose of study drug were excluded.
Time Frame: Extension study baseline, week 11 and week 28
Population: as for outcome 8
Measure: Median (Inter-Quartile Range); unit: mg/dl
Arm/Group | 20130356 SOC | 20130356 SOC + Cinacalcet | 20110100 SOC + Cinacalcet
Number analyzed (Participants) | 13 | 14 | 1
mg/dl
  Extension study baseline | 5.57 [4.86 to 6.19] | 6.05 [5.31 to 6.67] | 8.08 [8.08 to 8.08]
  Week 11: number analyzed (Participants) | 12 | 12 | 0
  Week 11 | 5.25 [4.55 to 5.80] | 6.20 [5.55 to 7.30] |
  Week 28: number analyzed (Participants) | 9 | 10 | 0
  Week 28 | 5.00 [4.30 to 5.60] | 5.95 [5.70 to 6.80] |

10. Secondary Outcome: Percentage of Participants Achieving ≥ 30% Reduction in iPTH From Day 1 of Cinacalcet Treatment to Mean Value During Weeks 11 and 15
Description: The percentage of participants who achieved ≥ 30% reduction in iPTH measured from the date the initial dose of cinacalcet was administered, in parent study 20130356 or 20110100 for participants who received cinacalcet in the parent study, or in the extension study for participants who received SOC only in parent study 20130356.
  Participants who had no iPTH values during weeks 11 and 15 were considered non-responders. Data collected more than 7 days after the last dose of study drug were excluded.
Time Frame: Baseline and weeks 11 and 15, relative to day 1 of cinacalcet treatment.
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 20130356 SOC | 20130356 SOC + Cinacalcet | 20110100 SOC + Cinacalcet
Number analyzed (Participants) | 13 | 14 | 1
percentage of participants | 30.8 [9.1 to 61.4] | 35.7 [12.8 to 64.9] | 100.0 [2.5 to 100.0]

11. Secondary Outcome: Percentage of Participants Achieving ≥ 30% Reduction in iPTH From Day 1 of Cinacalcet Treatment to Mean Value During Weeks 23 and 28
Description: The percentage of participants who achieved ≥ 30% reduction in iPTH measured from the date the initial dose of cinacalcet was administered, in parent study 20130356 or 20110100 for participants who received cinacalcet in the parent study, or in the extension study for participants who received SOC only in parent study 20130356.
  For participants who did not have an iPTH value during weeks 23 and 28, the mean of the last two available post-baseline values collected at protocol-specified visits was used. If only one post-baseline value was available, this single value was used. If no post-baseline value was available, the participant was considered a non-responder. Data collected more than 7 days after the last dose of study drug were excluded.
Time Frame: Baseline and weeks 23 and 28, relative to day 1 of cinacalcet treatment.
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 20130356 SOC | 20130356 SOC + Cinacalcet | 20110100 SOC + Cinacalcet
Number analyzed (Participants) | 13 | 14 | 1
percentage of participants | 23.1 [5.0 to 53.8] | 35.7 [12.8 to 64.9] | 0.0 [0.0 to 97.5]

12. Secondary Outcome: Percent Change From Day 1 of Cinacalcet Treatment in iPTH Over Time
Description: Percent change in iPTH measured from the date the initial dose of cinacalcet was administered, either in parent study 20130356 or 20110100, or in the extension study for participants who received SOC only in parent study 20130356.
  Data collected more than 7 days after the last dose of study drug were excluded.
Time Frame: Baseline and weeks 3, 7, 11, 15, 17, 18, 19, 20, 23, 27, 31, 35, 39, 43, 48, 52, relative to day 1 of cinacalcet treatment, and at the end of treatment visit and end of study visit (4 weeks after the end of treatment visit).
Population: as for outcome 8
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | 20130356 SOC | 20130356 SOC + Cinacalcet | 20110100 SOC + Cinacalcet
Number analyzed (Participants) | 13 | 14 | 1
percent change
  Week 3 | 10.16 [-4.42 to 20.24] | -6.88 [-30.86 to 41.81] | 55.54 [55.54 to 55.54]
  Week 7: number analyzed (Participants) | 13 | 13 | 1
  Week 7 | 1.99 [-37.82 to 17.42] | -4.96 [-40.93 to 32.44] | 9.78 [9.78 to 9.78]
  Week 11: number analyzed (Participants) | 12 | 13 | 1
  Week 11 | 19.75 [-27.88 to 84.96] | -7.64 [-30.77 to 13.37] | -7.00 [-7.00 to -7.00]
  Week 15: number analyzed (Participants) | 12 | 14 | 1
  Week 15 | -7.67 [-59.96 to 51.23] | -13.04 [-68.59 to 10.74] | -73.85 [-73.85 to -73.85]
  Week 17: number analyzed (Participants) | 2 | 12 | 1
  Week 17 | -23.93 [-59.61 to 11.75] | -3.09 [-40.52 to 21.40] | -20.02 [-20.02 to -20.02]
  Week 18: number analyzed (Participants) | 0 | 12 | 1
  Week 18 |  | -29.85 [-54.42 to 31.15] | -7.49 [-7.49 to -7.49]
  Week 19: number analyzed (Participants) | 10 | 12 | 0
  Week 19 | -37.17 [-69.24 to 21.47] | -3.50 [-50.02 to 19.16] |
  Week 20: number analyzed (Participants) | 1 | 11 | 1
  Week 20 | -13.12 [-13.12 to -13.12] | 0.44 [-35.10 to 66.13] | 160.80 [160.80 to 160.80]
  Week 23: number analyzed (Participants) | 10 | 14 | 0
  Week 23 | -9.05 [-52.43 to 28.64] | -6.65 [-35.13 to 83.11] |
  Week 27: number analyzed (Participants) | 10 | 13 | 0
  Week 27 | -8.50 [-69.20 to 18.78] | 16.36 [-59.79 to 50.23] |
  Week 31: number analyzed (Participants) | 0 | 13 | 0
  Week 31 |  | 32.30 [-58.73 to 75.48] |
  Week 35: number analyzed (Participants) | 0 | 12 | 0
  Week 35 |  | 16.82 [-70.15 to 82.83] |
  Week 39: number analyzed (Participants) | 0 | 12 | 0
  Week 39 |  | 0.09 [-58.27 to 86.94] |
  Week 43: number analyzed (Participants) | 0 | 12 | 0
  Week 43 |  | -17.13 [-47.15 to 47.30] |
  Week 48: number analyzed (Participants) | 0 | 10 | 0
  Week 48 |  | -45.67 [-66.01 to 33.64] |
  Week 52: number analyzed (Participants) | 0 | 1 | 0
  Week 52 |  | 86.50 [86.50 to 86.50] |
  End of treatment: number analyzed (Participants) | 10 | 12 | 0
  End of treatment | -8.50 [-69.20 to 18.78] | -45.67 [-74.62 to 34.62] |
  End of study: number analyzed (Participants) | 1 | 1 | 0
  End of study | 105.27 [105.27 to 105.27] | 20.21 [20.21 to 20.21] |

13. Secondary Outcome: Change From Day 1 of Cinacalcet Treatment in Serum Corrected Calcium Over Time
Description: Change in corrected calcium measured from the date the initial dose of cinacalcet was administered, either in parent study 20130356 or 20110100, or in the extension study for participants who received SOC only in parent study 20130356.
  Data collected more than 7 days after the last dose of study drug were excluded.
Time Frame: as for outcome 12
Population: as for outcome 8
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | 20130356 SOC | 20130356 SOC + Cinacalcet | 20110100 SOC + Cinacalcet
Number analyzed (Participants) | 13 | 14 | 1
mg/dL
  Week 3 | -0.18 [-0.26 to -0.11] | 0.19 [0.05 to 0.32] | -0.1 [-0.1 to -0.1]
  Week 7: number analyzed (Participants) | 13 | 13 | 1
  Week 7 | -0.34 [-0.44 to -0.24] | -0.01 [-0.23 to 0.21] | -0.5 [-0.5 to -0.5]
  Week 11: number analyzed (Participants) | 12 | 13 | 1
  Week 11 | -0.35 [-0.46 to -0.24] | -0.06 [-0.19 to 0.07] | -0.5 [-0.5 to -0.5]
  Week 15: number analyzed (Participants) | 12 | 14 | 1
  Week 15 | -0.37 [-0.62 to -0.12] | 0.06 [-0.18 to 0.30] | 0.5 [0.5 to 0.5]
  Week 17: number analyzed (Participants) | 2 | 12 | 1
  Week 17 | -0.02 [-0.24 to 0.20] | -0.11 [-0.45 to 0.22] | -0.8 [-0.8 to -0.8]
  Week 18: number analyzed (Participants) | 0 | 12 | 1
  Week 18 |  | -0.17 [-0.35 to 0.02] | -0.3 [-0.3 to -0.3]
  Week 19: number analyzed (Participants) | 10 | 12 | 1
  Week 19 | -0.43 [-0.60 to -0.26] | -0.20 [-0.37 to -0.03] | -0.1 [-0.1 to -0.1]
  Week 20: number analyzed (Participants) | 0 | 12 | 0
  Week 20 |  | -0.01 [-0.18 to 0.16] |
  Week 21: number analyzed (Participants) | 0 | 9 | 1
  Week 21 |  | -0.36 [-0.63 to -0.09] | -2.6 [-2.6 to -2.6]
  Week 23: number analyzed (Participants) | 9 | 12 | 0
  Week 23 | -0.18 [-0.24 to -0.12] | -0.20 [-0.47 to 0.08] |
  Week 27: number analyzed (Participants) | 9 | 13 | 0
  Week 27 | -0.14 [-0.25 to -0.02] | -0.24 [-0.41 to -0.07] |
  Week 31: number analyzed (Participants) | 0 | 13 | 0
  Week 31 |  | -0.00 [-0.20 to 0.19] |
  Week 35: number analyzed (Participants) | 0 | 12 | 0
  Week 35 |  | -0.42 [-0.57 to -0.26] |
  Week 39: number analyzed (Participants) | 0 | 12 | 0
  Week 39 |  | -0.63 [-0.84 to -0.43] |
  Week 43: number analyzed (Participants) | 0 | 12 | 0
  Week 43 |  | -0.37 [-0.63 to -0.11] |
  Week 48: number analyzed (Participants) | 0 | 10 | 0
  Week 48 |  | -0.55 [-0.87 to -0.23] |
  Week 52: number analyzed (Participants) | 0 | 1 | 0
  Week 52 |  | -0.16 [-0.16 to -0.16] |
  End of treatment: number analyzed (Participants) | 9 | 12 | 0
  End of treatment | 0.18 [0.02 to 0.34] | -0.04 [-0.26 to 0.18] |
  End of study: number analyzed (Participants) | 1 | 0 | 0
  End of study | 1.00 [1.00 to 1.00] |  |

14. Secondary Outcome: Change From Day 1 of Cinacalcet Treatment in Serum Phosphorus Over Time
Description: Change in phosphorus measured from the date the initial dose of cinacalcet was administered, either in parent study 20130356 or 20110100, or in the extension study for participants who received SOC only in parent study 20130356.
  Data collected more than 7 days after the last dose of study drug were excluded.
Time Frame: as for outcome 12
Population: as for outcome 8
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | 20130356 SOC | 20130356 SOC + Cinacalcet | 20110100 SOC + Cinacalcet
Number analyzed (Participants) | 13 | 14 | 1
mg/dL
  Week 3 | -0.24 [-0.56 to -0.08] | 0.81 [-0.54 to 1.07] | 5.6 [5.6 to 5.6]
  Week 7: number analyzed (Participants) | 13 | 13 | 1
  Week 7 | -0.16 [-0.50 to 0.17] | 0.37 [0.10 to 0.64] | 0.3 [0.3 to 0.3]
  Week 11: number analyzed (Participants) | 12 | 12 | 1
  Week 11 | 0.01 [-0.33 to 0.36] | 1.17 [0.87 to 1.47] | 0 [0 to 0]
  Week 15: number analyzed (Participants) | 12 | 14 | 1
  Week 15 | -0.52 [-0.79 to -0.25] | 0.96 [0.71 to 1.20] | -1.9 [-1.9 to -1.9]
  Week 17: number analyzed (Participants) | 2 | 12 | 0
  Week 17 | -0.08 [-0.19 to 0.03] | 1.57 [0.96 to 2.19] |
  Week 18: number analyzed (Participants) | 0 | 12 | 1
  Week 18 |  | 0.61 [0.30 to 0.93] | -0.9 [-0.9 to -0.9]
  Week 19: number analyzed (Participants) | 10 | 12 | 1
  Week 19 | -0.45 [-0.74 to -0.16] | 0.91 [0.37 to 1.44] | -0.3 [-0.3 to -0.3]
  Week 20: number analyzed (Participants) | 0 | 11 | 0
  Week 20 |  | 0.84 [0.16 to 1.51] |
  Week 21: number analyzed (Participants) | 0 | 9 | 1
  Week 21 |  | 0.17 [-0.67 to 1.01] | 0.1 [0.1 to 0.1]
  Week 23: number analyzed (Participants) | 9 | 12 | 0
  Week 23 | -0.37 [-0.78 to 0.05] | 0.55 [0.12 to 0.98] |
  Week 27: number analyzed (Participants) | 9 | 13 | 0
  Week 27 | -0.18 [-0.53 to 0.18] | 0.76 [0.27 to 1.24] |
  Week 31: number analyzed (Participants) | 0 | 13 | 0
  Week 31 |  | 0.83 [0.24 to 1.42] |
  Week 35: number analyzed (Participants) | 0 | 12 | 0
  Week 35 |  | -0.03 [-0.51 to 0.45] |
  Week 39: number analyzed (Participants) | 0 | 12 | 0
  Week 39 |  | 0.40 [-0.11 to 0.91] |
  Week 43: number analyzed (Participants) | 0 | 12 | 0
  Week 43 |  | 0.33 [-0.21 to 0.86] |
  Week 48: number analyzed (Participants) | 0 | 8 | 0
  Week 48 |  | 0.60 [-0.21 to 1.42] |
  Week 52: number analyzed (Participants) | 0 | 1 | 0
  Week 52 |  | 0.61 [0.61 to 0.61] |
  End of treatment: number analyzed (Participants) | 9 | 10 | 0
  End of treatment | -0.18 [-0.53 to 0.18] | 0.43 [-0.25 to 1.11] |
  End of study: number analyzed (Participants) | 1 | 0 | 0
  End of study | 1.20 [1.20 to 1.20] |  |

ADVERSE EVENTS:
Time Frame: From first dose of study drug in the extension study up to 4 weeks after the last dose; 32 weeks.
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Groups:
- Total: All participants who received cinacalcet in study 20140159.
Arm/Group | 20130356 SOC | 20130356 SOC + Cinacalcet | 20110100 SOC + Cinacalcet | Total
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/14 | 1/1 | 1/28
Serious Adverse Events (participants affected / at risk) | 2/13 | 6/14 | 1/1 | 9/28
Other Adverse Events (participants affected / at risk) | 9/13 | 10/14 | 1/1 | 20/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 20130356 SOC (N=13) | 20130356 SOC + Cinacalcet (N=14) | 20110100 SOC + Cinacalcet (N=1) | Total (N=28)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Goitre (Endocrine disorders) | 1 | 0 | 0 | 1
Gastroduodenitis (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Fatigue (General disorders) | 0 | 1 | 0 | 1
Local swelling (General disorders) | 0 | 1 | 0 | 1
Pyrexia (General disorders) | 0 | 1 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 1
Device related infection (Infections and infestations) | 0 | 2 | 0 | 2
Pericarditis infective (Infections and infestations) | 0 | 1 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 1
Staphylococcal infection (Infections and infestations) | 0 | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 1
Device damage (Product Issues) | 0 | 1 | 0 | 1
Device dislocation (Product Issues) | 0 | 1 | 1 | 2
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Catheter placement (Surgical and medical procedures) | 0 | 1 | 0 | 1
Venous occlusion (Vascular disorders) | 0 | 1 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 20130356 SOC (N=13) | 20130356 SOC + Cinacalcet (N=14) | 20110100 SOC + Cinacalcet (N=1) | Total (N=28)
Left ventricular hypertrophy (Cardiac disorders) | 0 | 1 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 1
Goitre (Endocrine disorders) | 1 | 0 | 0 | 1
Hyperparathyroidism secondary (Endocrine disorders) | 0 | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 1 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Duodenogastric reflux (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Gastritis erosive (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Gastroduodenitis (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2 | 0 | 2
Chest pain (General disorders) | 1 | 1 | 0 | 2
Complication associated with device (General disorders) | 0 | 1 | 0 | 1
Local swelling (General disorders) | 0 | 1 | 0 | 1
Mass (General disorders) | 1 | 0 | 0 | 1
Nodule (General disorders) | 0 | 1 | 0 | 1
Peripheral swelling (General disorders) | 0 | 1 | 0 | 1
Pyrexia (General disorders) | 0 | 2 | 0 | 2
Hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 1
Herpes virus infection (Infections and infestations) | 1 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 1 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 2 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 1
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Heat exhaustion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Ulna fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Adjusted calcium decreased (Investigations) | 1 | 1 | 0 | 2
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 0 | 1
Blood calcium decreased (Investigations) | 1 | 1 | 0 | 2
Blood parathyroid hormone decreased (Investigations) | 1 | 0 | 0 | 1
C-reactive protein increased (Investigations) | 0 | 1 | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 1 | 0 | 1
Red blood cell sedimentation rate increased (Investigations) | 0 | 1 | 0 | 1
Weight decreased (Investigations) | 0 | 1 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 0 | 1
Loss of consciousness (Nervous system disorders) | 0 | 1 | 0 | 1
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 1
Tremor (Nervous system disorders) | 1 | 0 | 0 | 1
Major depression (Psychiatric disorders) | 0 | 1 | 0 | 1
Staring (Psychiatric disorders) | 0 | 1 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Pulmonary calcification (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Catheter placement (Surgical and medical procedures) | 0 | 1 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 1 | 1
Venous haemorrhage (Vascular disorders) | 1 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2017-08-21): https://cdn.clinicaltrials.gov/large-docs/17/NCT02341417/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-21): https://cdn.clinicaltrials.gov/large-docs/17/NCT02341417/SAP_001.pdf